CLINICAL TRIAL: NCT06467903
Title: A Prospective, Comparative Multicenter Evaluation Conducted to Capture Patients With Diabetic Retinopathy in General Practitioners, Using the SW as Medical Device and the SW as MD Comparator, When Evaluating the Patient's Retinal Image
Brief Title: Evaluation Conducted to Capture Patients With Diabetic Retinopathy in General Practitioners, Using SW as Medical Device
Acronym: Retina
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bonmedix Holding a.s. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Retina_01_2024; sukls117945/2024 (Other: SUKL)
Record Dates: First submitted 2024-06-10; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: specific screening exhamination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm - 1000 patients, DR screening (Experimental): SW as medical devices(investigational device) to evaluate the retinal image of the patient's eye (to identify if the patient has DR or if the patient is healthy) .
  Interventions: Device: SW as medical devices(comperator) to evaluate the retinal image of the patient's eye (to identify if the patient has DR or if the patient is healthy) .

INTERVENTIONS:
Device: SW as medical devices(comperator) to evaluate the retinal image of the patient's eye (to identify if the patient has DR or if the patient is healthy) . — second AI medical device to evaluate the retinal image of the patient's eye. two AI as MD will be evaluating the retinal image

SUMMARY:
A prospective, comparative multicenter evaluation conducted to capture patients with diabetic retinopathy in general practitioners, using AI medical device

DETAILED DESCRIPTION:
A prospective, comparative multicenter evaluation conducted to capture patients with diabetic retinopathy in general practitioners, using the SWaMD medical device and the SWaMD comparator, when evaluating the patients retinal image

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 40 years
* Signed informed consent
* Confirmed type 1 or 2 diabetes mellitus

Exclusion Criteria:

* Ocular findings that do not allow retinal photography (significant nystagmus, corneal leukoma, dense cataract, hemophthalmus, etc.)
* Patient has a condition or is in a situation that, in the opinion of the investigator, may bias the results of the study, may significantly interfere with the patient's participation in the investigation, or may result in unproducible photographs of a dilated ocular fundus
* Patients with restrictions on personal freedom by administrative or legal order

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-10-28 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | 3 months
  The sensitivity and specificity will be calculated using the evaluation of independent masked expert (ophthalmologist) as gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Šonka, MD, Principal Investigator — GP
Locations (1):
- Jakub Sedivy, Příbram, Or, Czechia

IPD SHARING:
Plan to Share IPD: No